CLINICAL TRIAL: NCT04659889
Title: Analysis of the Relationship Between Clinical and Haematological Phenotypes in Long COVID
Brief Title: Clinical and Haematological Phenotypes in Long COVID
Status: Completed | Type: Observational
Sponsor: HCA International Limited (Other)
Responsible Party: Principal Investigator, Dr Paul Glynne, Consultant Physician, HCA International Limited
Other Study IDs: LCV
Record Dates: First submitted 2020-12-07; First posted 2020-12-09 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Long Covid; Covid19
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; COVID-19 | interventions — Blood Specimen Collection; Phlebotomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with clinical features of Long Covid: Patients who have had COVID-19 (PCR proven and/or clinical features of COVID-19) who are currently displaying symptoms of long Covid
  Interventions: Diagnostic Test: Blood sampling (venesection)
- Patients with no symptoms of Long Covid: Patients who have had COVID-19 (PCR proven and/or clinical features of COVID-19) who are not displaying symptoms of long Covid
  Interventions: Diagnostic Test: Blood sampling (venesection)

INTERVENTIONS:
Diagnostic Test: Blood sampling (venesection) — All study participants will have a single blood test to analyse the following parameters:
  (i) Serum biochemistry, CRP, Thyroid function and liver enzymes (ii) FBC, d-Dimer, ESR, Blood film (iii) SARS-CoV2 antibody status and serum save (iv) Peripheral blood immunophenotyping.

SUMMARY:
Analysis of the relationship between clinical characteristics and haematological parameters in long COVID.

The novel coronavirus (Covid19) pandemic declared by the World Health Organisation in March 2020 has had an enormous huge impact upon health, health systems and society. Early research has focused on the acute illness caused by the virus. It is now clear that significant numbers of patients infected with Covid19 continue to suffer with multiple, often severe, unexplained symptoms for months after initial infection, so-called long-Covid.

Long-Covid symptoms are typically multi-system in their presentation comprising constitutional changes (e.g. fever and fatigue), neuropsychiatric disturbance (e.g. anxiety, insomnia and brain fog), neurosensory symptoms (e.g. headaches and pins and needles), cardiorespiratory effects (e.g. breathlessness and chest pain), gastrointestinal dysfunction (e.g. diarrhoea and food intolerances) and dermatological changes (e.g. rashes and vascular changes).

The objectives of this observational, cross-sectional, case-control study are to describe long-Covid clinical phenotypes and to explore whether clinical symptom presentations correlate with haematological and other inflammatory blood abnormalities that might shed insight into underlying pathogenic mechanisms.

The study will require the participation of long-Covid patients, seen in an outpatient setting at The Physicians' Clinic, and will correlate clinical symptom phenotypes with laboratory parameters we believe might be relevant to long-Covid. Recruitment of asymptomatic patients, who have recovered from Covid19 infection, will provide a control patient group. Eligible patients will be sent a patient information sheet, describing the study objectives and protocol, inviting them to participate in the study and seeking consent for their participation, which will require analysis of their [anonymised] clinical and laboratory data. Clinical information will be retrieved from patient case records and patients will be asked to complete a symptom questionnaire. All patients will require one blood sample to be taken which will typically form part of their clinical care. Recruitment will occur over a 6 month period.

DETAILED DESCRIPTION:
There are estimated to be tens of thousands of long-Covid patients in the UK, and the number is set to grow as the pandemic continues. Little is known about the cause of long-Covid clinical syndromes and there are no evidence-based treatments available to patients. There is therefore an urgent need to undertake research into long-Covid.

Long-Covid referral to our general medical outpatient clinics has been growing, as these patients typically present with multiple symptoms that require a holistic approach to patient care. Patients are often distressed and disabled by their symptoms, exacerbated by the lack of any detailed understanding about their condition, and the absence of specific treatment strategies. Anecdotal reports of ongoing inflammation in long-Covid, not typically measurable in routine blood tests, have prompted interest in exploring the nature of this inflammation further. In addition, some long-Covid patients have reported clinical improvement following empiric treatment with anti-inflammatory medications including anti-histamines and corticosteroids. These clinical observations, and the enthusiasm expressed by the long-Covid patient community for further research to be conducted, have been the key drivers for this study. Patients attending our clinics have all without exception expressed their interest in participating in this work.

This small sample size study sets out to explore whether there are identifiable abnormalities in the blood cells of long-Covid patients that might correlate with patients' clinical presentations which may in turn trigger further avenues of investigation.

The study participants are all patients with a history of Covid19 infection and who either have ongoing symptoms or who have fully recovered. The clinical information is available in case records as part clinical care and patients' blood samples are sent for analysis as part of ongoing clinical care. Patients are informed about their blood test results as part of ongoing clinic care. All patients are provided with information about the study and asked to consent to their anonymised clinical and laboratory data being used as part of this observational study. We also seek consent to save serum for additional blood analysis depending on the results of the initial study. No genetic investigations will be conducted.

This study does not involve any treatment intervention, and there is no risk of harm to patients. The use of person-identifiable information will be restricted to an absolute minimum, and all data will be anonymised for purposes of our study analysis. The members of the research team all work within one organisation adhering to GDPR standards, and all email communication remains within that organisation and is password-protected. No conflicts of interest have been identified. We have undertaken to share individual results with participating patients by the end of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients post documented SARS-CoV-2 infection displaying symptoms of long Covid
2. Asymptomatic post documented SARS-CoV-2 infection
3. All patients will be aged 18 or over

Exclusion Criteria:

1. Patients below the age of 18
2. Patients who have not previously had COVID-19
3. Any adult deemed to trigger consideration of being a Vulnerable Adult.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The first group will be patients post documented SARS-CoV-2 infection displaying symptoms of long Covid and the second group will be patients who are asymptomatic post documented SARS-CoV-2 infection
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Observation of frequency of abnormal haematological parameters and association with long-Covid clinical phenotypes versus controls. | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- The Physicians' Clinic, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No